CLINICAL TRIAL: NCT01020500
Title: An International, Prospective Cohort to Document the Effectiveness of One BoNT-A Injection Cycle Based on Attainment of Individual Person-centred Goals in Adult Subjects Suffering From Upper Limb Spasticity Following Stroke
Brief Title: To Document the Effectiveness of BoNT-A Injection in Adult Subjects With Upper Limb Spasticity Following Stroke
Acronym: ULIS2
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-79-52120-138
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to assess the responder rate as defined by the achievement of the primary goal from the Goal Attainment Scale following one BoNT-A injection cycle in accordance with routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb spasticity following stroke
* At least a 12-week interval between the last injection (BoNT-A or BoNT-B) and inclusion
* Decision already been agreed to inject BoNT-A
* Agreement with the subject on goal setting

Exclusion Criteria:

* Contraindications to any BoNT-A preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Clinics
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Responder rate as defined by the achievement of the primary goal from the Goal Attainment Scale (GAS) following one BoNT-A injection cycle in accordance with routine practices | Around 3 to 5 months post injection

SECONDARY OUTCOMES:
Overall attainment of the treatment goals using the GAS T score | Around 3 to 5 months post injection
Result of standardized outcome measures (e.g., muscle tone reduction, pain scores, arm function test) | Around 3 to 5 months post injection
Global assessment of benefits by both the investigator and the subject (or guardian) | Around 3 to 5 months post injection

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (96):
- Australia (6):
  - Rankin Park (site 036006), Newcastle
  - Northshore Private Hospital (site 036003), Sydney
  - Royal Prince Alfred Hospital (site 036005), Sydney
  - Ryde Rehabilitation Center (site 036002), Sydney
  - St Joseph's Hospital (site 036004), Sydney
  - St Vincent's Hospital (site 036001), Sydney
- Austria (2):
  - NÖ LKH Grimmenstein-Hochegg (site 040002), Grimmenstein
  - Gaital-Kliniken Hermagor (site 040001), Hermagor
- Belgium (4):
  - Revalidatieziekenhuis Hof ter Schelde, August Vermeylenlaan 6 (site 056001), Antwerp
  - AZ St. Jan, Ruddershove 10, (site 056002), Bruges
  - UCL St. Luc Département de médecine, physique et de readaptation motrice, Avenue Hippocrate 10 (site 056004), Brussels
  - Cliniques Universitaires UCL de Mont-Godinne, Avenue Dr. G. Therasse (site 056003), Yvoir
- Rehabilitation Unit, Tung Wah Hospital, 12 Po Yan Street, Sheung Wan (site 344001), Hong Kong, China
- Czechia (2):
  - Faculty Hospital Brno (site 203002), Brno
  - Hospital Pardubice, Neurology dept. (site 203001), Pardubice
- Denmark (3):
  - Aarhus University Hospital, Neurolog avd.F-NEU-Cent (Site 208001), Aarhus
  - Herlev Hospital, Herlev Ringvej (Site 208004), Copenhagen
  - Neurologisk afdeling N, Amtssygehuset i Glostrup (Site 208003), Glostrup Municipality
- Finland (3):
  - Department of Physical and Rehabilitation Medicine/Central Hospital of Central Finland (Site 246005), Jyväskylä
  - Invalidförbundets Rehabiliteringscenter i Lappland (Site 246004), Rovaniemi
  - Neurologiska Polikliniken, Tampere University Hospital (site 246001), Tampere
- France (19):
  - Centre Régional de Rééducation et Réadaptation fonctionnelle (site 250008), Angers
  - Centre de Rééducation Fonctionnelle du Mont Veyrier Rééducation fonctionnelle (site 250021), Argonay
  - Hôpital Jean Minjoz/Méd.physique réadaptation (site 250016), Besançon
  - Hôpital Pellegrin/Rééducation fonctionnelle (site 250012), Bordeaux
  - Centre Médecine Physique Réadaptation/Rééducation Neurologique (site 250013), Coubert
  - Hopital Albert Chenevier/Neurologie, (site 250010), Créteil
  - CHU Hôpital SUD/Institut de Rééducation (site 250007), Échirolles
  - Hôpital Raymond Poincaré/Rééducation neurologique (site 250002), Garches
  - CHRU Lille/Rééducation Neurologique (site 250018), Lille
  - Hopital Jean Rebeyrol/Médecine Physique et de Réadaptation (site 250006), Limoges
  - Centre Médico-Chirurgical de Réadaptation des Massues (Site 250005), Lyon
  - Hôpital Timone Adultes/Rééducation fonctionnelle (site 250020), Marseille
  - CHU Lapeyronie /Rééducation fonctionnelle (site 250014), Montpellier
  - CHU de Nantes/Médecine physique et de réadaptation neurologique (site 250017), Nantes
  - Médecine Physique et de Réadaptation Fondation Hospitalière Sainte Marie (site 250001), Paris
  - Hôpital Sébastopol/Rééducation Fonctionnelle (site 250004), Reims
  - Hôpital Pontchaillou/Rééducation Fonctionnelle (site 250003), Rennes
  - Hôpital Hautepierre/Rééducation fonctionnellev (site 250011), Strasbourg
  - Hôpital Rangueil/Médecine Physique réadaptation (site 250015), Toulouse
- Germany (7):
  - Sächs. KH Neurologie, Hufelandstr. 15 (site 276006), Arnsdorf
  - Kinik für Neurologie Paracelsusring 6a (site 276003), Beelitz
  - NRZ Neurologisches Rehazentrum (site 276004) Muldentalweg 1, Bennewitz
  - Praxis für Neurologie, Dalberger Str. 6 (site 276007), Frankfurt
  - Kliniken der Medizinischen Hochschule (Neurologische Klinik), Carl-Neuberg-Str. 1 (site 276005), Hanover
  - Praxis für Neurologie Mittelstr. 4 (site 276008), Mannheim
  - Paracelsus Klinik Werdauer Str. 68 (site 276002), Zwickau
- Italy (6):
  - Clinica di Neuroriabilitatione - Az. Osp. Univ. Ospedali Riuniti (site 380004), Ancona
  - Azienda Ospedaliera Universitaria (site 380012), Ferrara
  - Ospedale Valduce, Costa Masnaga (site 380001), Lecco
  - Laboratorio analisi del Movimento U.O.R.R.F. -Ospedale Santa Corona (site 380002), Pietra Ligure
  - Ospedale Cisanello (site 380010), Pisa
  - Ospedale S. Bartolomeo (site 380005), Sarzana
- Malaysia (2):
  - Hospital Kuala Lumpur (site 458002), Kuala Lumpur
  - Universiti Malaya Medical Center/Department of Neurology / Department of Rehabilitation Medicine (site 458001), Kuala Lumpur
- Mexico (2):
  - Colonia Ladrón de Guevara (Site 484001), Guadalajara, Jalisco
  - Angeles del Pedregal (Site 484002), México
- Philippines (2):
  - Perpetual Succour Hospital (site 608002), Cebu City
  - Metropolitan Medical Center (site 608001), Manila
- Portugal (5):
  - Centro de Medicina de Reabilitação de Alcoitão (site 620001), Alcabideche
  - Centro Hospitalar de Coimbra - Quinta dos Vales (site 620005), Coimbra
  - Hospital Distrital de Faro (site 620004), Faro
  - Hospital Egas Moniz, Centro Hospitalar Lisboa Ocidental (site 620003), Lisbon
  - Hospital Geral de Santo Antonio, Centro Hospitalar do Porto (site 620002), Porto
- Russia (7):
  - Municipal health care institution "City clinical hospital #3" (site 643006), Chelyabinsk
  - State Institution "Interregional clinical diagnostic centre" (site 643002), Kazan'
  - Municipal health care institution "City hospital #2 "Krasnodar Multidisciplinary medical diagnostic association" (site 643004), Krasnodar
  - State Educational Institution of high professional education "Krasnoyarsk State Medical Academy of Roszdrav" (site 643007), Krasnoyarsk
  - Federal State Institution "Medical Rehabilitation Centre of Roszdrav" (site 643001), Moscow
  - State Novosibirsk Regional Clinical Diagnostic Centre (site 643005), Novosibirsk
  - State Educational Institution of high professional education "St-Peterbusrg state medical university named after I.P. Pavlov of Roszdrav" (site 643003), St-Peterburg
- Singapore (2):
  - Singapore General Hospital, Department of Rehabilitation Medicine (site 702002), Singapore
  - Tan Tock Seng Hospital/TTSH Rehabilitation Centre (site 702001), Singapore
- South Korea (6):
  - Catholic University Daejeon St. Mary's Hospital, Daeheung-dong, Jung-gu, (site 410004), Daejeon
  - Inha University Hospital, #7-206 Shinheungdong-ga,Jjung-gu (site 410006), Incheon
  - Samsung Medical Center, #50 Ilwon-dong, Gangnam-gu (site 410002), Seoul
  - Dept. for Rehabilitation Asan Medical Center (site 410005), Seoul
  - Dept. of Rehabilitation Seoul National University Bundang Hospital (site 410003), Seoul
  - Dept. of Rehabilitation Yonsei University Severance Hospital (site 410001), Seoul
- Spain (4):
  - Hospital La Paz / Servicio de Rehabilitación (site 724006), Madrid
  - Hospital Morales Meseguer / Servicio de Rehabilitación (site 724005), Murcia
  - Hospital Marqués de Valdecilla/ Servicio de Rehabilitación (site 724009), Santander
  - Hospital Universitario La Fe (Site 724003), Valencia
- Sweden (4):
  - Mälarsjukhuset, Dept. Of Neurology (site 752001), Eskilstuna
  - Dept. Of Neurology, Nyköping Hospital (site 752002), Nyköping
  - Östersunds Rehab Centrum (site 752004), Östersund
  - Läkarhuset Odenplan, Neuro Unit (site 752003), Stockholm
- Taiwan (2):
  - China Medical University Hospital, Department of Physical Medicine & Rehabilitation (site 158002), Taichung
  - Veteran General Hospital (site 158001), Taipei
- Thailand (2):
  - King Chulalongkorn Memorial Hospital/Department of Rehabilitation Medicine (site 764002), Bangkok
  - Siriraj Hospital/Department of Rehabilitation Medicine (site 764001), Bangkok
- United Kingdom (5):
  - Dewsbury District Hospital (site 826004), Dewsbury
  - Medway Maritime Hospital (site 826002), Gillingham
  - Lincoln County Hospital (site 826001), Lincoln
  - Regional Rehabilitation Unit, Northwick Park Hospital (site 826006), Middlesex
  - West Midlands/Rehabilitation Centre (826005), Plymouth

REFERENCES:
- [Derived] Fheodoroff K, Ashford S, Jacinto J, Maisonobe P, Balcaitiene J, Turner-Stokes L. Factors influencing goal attainment in patients with post-stroke upper limb spasticity following treatment with botulinum toxin A in real-life clinical practice: sub-analyses from the Upper Limb International Spasticity (ULIS)-II Study. Toxins (Basel). 2015 Apr 8;7(4):1192-205. doi: 10.3390/toxins7041192. PMID 25856546
- [Derived] Turner-Stokes L, Fheodoroff K, Jacinto J, Maisonobe P. Results from the Upper Limb International Spasticity Study-II (ULISII):a large, international, prospective cohort study investigating practice and goal attainment following treatment with botulinum toxin A in real-life clinical management. BMJ Open. 2013 Jun 20;3(6):e002771. doi: 10.1136/bmjopen-2013-002771. PMID 23794582
- [Derived] Turner-Stokes L, Fheodoroff K, Jacinto J, Maisonobe P, Zakine B. Upper limb international spasticity study: rationale and protocol for a large, international, multicentre prospective cohort study investigating management and goal attainment following treatment with botulinum toxin A in real-life clinical practice. BMJ Open. 2013 Mar 18;3(3):e002230. doi: 10.1136/bmjopen-2012-002230. PMID 23512837